CLINICAL TRIAL: NCT05194202
Title: Promoting Healthy Relationships Among At-Risk Adolescents: A Feasibility Trial in the Emergency Department
Brief Title: Emergency Department Healthcare Education Assessment and Response for Teen Relationships: A Pilot Feasibility Study
Acronym: ED-HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kimberly Randell, Physician, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00001967; K23HD098299 (NIH)
Record Dates: First submitted 2021-10-18; First posted 2022-01-18 (Actual); Results first posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Behavior; Emergency Department; Abuse Physical; Abuse Mental; Abuse Verbal; Abuse Domestic; HEART; Intimate Partner Violence
MeSH Terms: conditions — Adolescent Behavior; Emergencies

STUDY DESIGN:
Intervention Model Description: Adolescents will be enrolled in one of two arms: Emergency Department Healthcare Education Assessment and Response for Teen Relationships (ED-HEART) (intervention arm) or Enhanced Usual Care (control arm). Adolescents will complete study surveys at baseline (Baseline Survey; intervention and control arms), immediately post-intervention (Exit Survey, intervention arm), and 12 weeks after intervention delivery (Follow-up Survey, intervention and control arms).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ED-HEART (Intervention Arm) (Experimental): All adolescents take a baseline survey in the Emergency Department (ED), receive Emergency Department Healthcare Education Assessment and Response for Teen Relationships (ED HEART) by a trained health educator, complete an exit survey while in the ED, complete a 6-week check-in to confirm contact information and aid retention, and complete a 12-week follow up survey.
  Interventions: Behavioral: ED-HEART
- Enhanced Standard Care (Control Arm) (No Intervention): All adolescents take a baseline survey in the Emergency Department (ED), receive enhanced standard care (i.e., standard care + teen resource list), complete a 6-week check in to confirm contact information and aid retention, and complete a 12-week follow up survey.

INTERVENTIONS:
Behavioral: ED-HEART — Behavioral intervention that assesses 1) healthy and unhealthy relationship behaviors, 2) conversation with partners around boundaries within relationships, 3) harm reduction strategies, and 4) resources for Adolescent Relationship Abuse (ARA) and related concerns, including Point of Care (POC) Reproductive and Sexual Health (RSH) harm reduction resources.
  Arms: ED-HEART (Intervention Arm)

SUMMARY:
This is a single-site, randomized, controlled trial. Investigators will evaluate feasibility of the Emergency Department Healthcare Education Assessment and Response for Teen Relationships (ED-HEART) intervention among adolescents age 14-19 years receiving care in the Children's Mercy emergency department.

DETAILED DESCRIPTION:
This study is a mixed methods feasibility evaluation that will use a randomized controlled trial to assess feasibility of Emergency Department Healthcare Education Assessment and Response for Teen Relationships (ED-HEART) (intervention arm: ED-HEART + teen resource list; control arm: enhanced standard care [standard care + teen resource list]). Adolescents age 14-19 years will be recruited and enrolled during an emergency department visit. Investigators will evaluate feasibility using the eight Bowen model feasibility constructs: acceptability, demand, implementation, practicality, adaptation, integration, expansion, and limited-efficacy testing. Investigators will also examine theory of planned behavior constructs (attitudes, beliefs, perceived behavioral control, intention) to facilitate exploratory analysis of factors that may contribute to differential outcomes.

ELIGIBILITY:
Inclusion Criteria:

* emergency department (ED) patient 14-19 years of age.

Exclusion Criteria:

* Developmental delay, severe illness, or cognitive impairment precluding informed consent/assent or completion of study activities, as determined by ED team or study team.
* Current ED evaluation for acute sexual assault/abuse.
* Current mental or behavioral health symptoms precluding completion of study activities, as determined by ED team or study team.
* Caregiver declines to step out to allow assent/consent in private or adolescent declines for caregiver to step out to allow assent/consent or participation in private.
* Adolescent is non-English speaking.
* Parent is non-English or non-Spanish speaking.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Study information will be shared with other members on the research team. Study data will be collected and stored via the Research Electronic Data Capture (REDCap) system. De-identifiable information may also be shared with other researchers.
Supporting Information: SAP
Time Frame: 12 months after study completion; indefinitely
Access Criteria: Researchers should contact the PI (Randell) with any requests for use of the data

RESULTS

PARTICIPANT FLOW:
Groups:
- ED-HEART (Intervention Arm): All adolescents take a baseline survey in the Emergency Department (ED), receive Emergency Department Healthcare Education Assessment and Response for Teen Relationships (ED HEART) by a trained health educator, complete an exit survey while in the ED, complete a 6-week check-in to confirm contact information and aid retention, and complete a 12-week follow up survey.
  ED-HEART: Behavioral intervention that addresses 1) healthy and unhealthy relationship behaviors, 2) conversation with partners around boundaries within relationships, 3) harm reduction strategies, and 4) resources for Adolescent Relationship Abuse (ARA) and related concerns, including Point of Care (POC) Reproductive and Sexual Health (RSH) harm reduction resources.
Period: Overall Study
Arm/Group | ED-HEART (Intervention Arm) | Enhanced Standard Care (Control Arm)
Started | 88 | 87
Completed | 39 | 39
Not Completed | 49 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ED-HEART (Intervention Arm) | Enhanced Standard Care (Control Arm) | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (1.5) | 15.7 (1.3) | 15.9 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 38 | 36 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 26 | 52
  Not Hispanic or Latino | 62 | 60 | 122
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 24 | 28 | 52
  White | 38 | 34 | 72
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  United States | 88 | 87 | 175
Commercial Insurance [Count of Participants; unit: Participants] | 24 | 31 | 55
History of adolescent relationship abuse [Count of Participants; unit: Participants] — Report of ARA victimization will be considered positive for any positive answer to one or more of six survey items assessing physical ARA, sexual ARA, sexual exploitation within a dating relationship, and (among females) reproductive coercion.
  Participants | 15 | 16 | 31
History of dating [Count of Participants; unit: Participants]
  History of dating | 76 | 72 | 148
  No history of dating | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Participant Acceptability Ratings for Healthcare Provider Discussions on Relationships in ED-Heart Intervention Arm
Description: 1 survey item (investigator-developed) on acceptability of healthcare providers discussing healthy/unhealthy relationships, rated using 5-point Likert scale (strongly disagree/1 to strongly agree/5)
Time Frame: 12 weeks
Population: Intervention participants answering acceptability item 1 on follow up survey
Measure: Count of Participants; unit: Participants
Arm/Group | ED-HEART (Intervention Arm)
Number analyzed (Participants) | 45
Participants
  Strongly agree/agree | 39
  Strongly disagree/disagree/neutral | 6
Statistical Analysis 1: Comparison: ED-HEART (Intervention Arm); Our null hypothesis for the acceptability was P0 great than or equal to 85% vs. the alternative P0 less than 85%. Acceptability responses were dichotomized to include neutral with strongly disagree/disagree; Test type: Other; p = .622, one-sample test of proportions; Hypothesis was evaluated using a one-tailed, one-proportion z-test

2. Primary Outcome: Participant Acceptability Ratings for ED-based Relationship Intervention in ED-Heart Intervention Arm
Description: 1 survey item (investigator-developed) on acceptability of emergency department based healthy/unhealthy relationships intervention, rated using 5-point Likert scale (strongly disagree/1 to strongly agree/5)
Time Frame: 12 weeks
Population: Intervention participants answering follow up survey acceptability of ED-based adolescent relationship intervention
Measure: Count of Participants; unit: Participants
Arm/Group | ED-HEART (Intervention Arm)
Number analyzed (Participants) | 45
Participants
  Strongly agree/agree | 34
  Strongly disagree/disagree/neutral | 11
Statistical Analysis 1: Comparison: ED-HEART (Intervention Arm); Our null hypothesis for the acceptabnility of the ED-Heart was P0 great than or equal to 85% vs. the alternative P0 less than 85%. Acceptability responses were dichotomized to include neutral with strongly disagree/disagree; Test type: Other; p = .038, one sample test of proportions; Hypothesis was evaluated using a one-tailed, one-proportion z-test

3. Secondary Outcome: ARA Victimization
Description: Report of ARA victimization will be considered positive for any positive answer to one or more of six survey items assessing physical ARA, sexual ARA, sexual exploitation within a dating relationship, and (among females) reproductive coercion.
Time Frame: 12 weeks
Population: Intervention and control arm participants who completed follow up surveys
Measure: Count of Participants; unit: Participants
Arm/Group | ED-HEART (Intervention Arm) | Enhanced Standard Care (Control Arm)
Number analyzed (Participants) | 47 | 54
Participants | 1 | 5

4. Secondary Outcome: Recognition of Abusive Behaviors
Description: 19 survey items, adapted from the Recognition of ARA Scale. Each item answered with 5-point Likert scale that categorizes each behavior from not abusive (1) to extremely abusive (5). Scored as mean; higher score indicates increased recognition of behaviors as abusive.
Time Frame: 12 weeks
Population: Intervention and control arm participants who completed follow up surveys
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ED-HEART (Intervention Arm) | Enhanced Standard Care (Control Arm)
Number analyzed (Participants) | 47 | 54
score on a scale | 4.18 (0.66) | 4.26 (0.54)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Definitions do not differ from clinicaltrials.gov definitions.
Arm/Group | ED-HEART (Intervention Arm) | Enhanced Standard Care (Control Arm)
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/87
Other Adverse Events (participants affected / at risk) | 0/88 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/02/NCT05194202/Prot_001.pdf
  • Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05194202/SAP_002.pdf
  • Informed Consent Form (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT05194202/ICF_000.pdf